CLINICAL TRIAL: NCT02513017
Title: Insomnia and Cardiovascular Diseases: Influence of Behavioral Treatments and Preferences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Souraya Sidani, Professor and Canada Research Chair, Toronto Metropolitan University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PCR - 101411
Record Dates: First submitted 2015-07-22; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Insomnia; Cardiovascular Disease
Keywords: partially randomized clinical trial; cardiovascular disease; insomnia; preference; acceptability
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stimulus Control Instructions (SCI) (Experimental): SCI is a behavioral treatment that aims to assist persons with insomnia to re-associate the bed and the bedroom with falling asleep or back to sleep, and to acquire a consistent sleep pattern. SCI entails specific instructions that focus on developing new sleep habits, such as avoiding activities other than sleep (e.g., reading, watching TV) in bed, and getting out of bed if unable to fall asleep and engaging in quiet activities until sleepy.
  A trained therapist will deliver the session in which the following topics will be covered: education about sleep, factors that influence sleep, behaviors that promote or interfere with sleep, and SCI. The session will be offered in a small group (4-6) format, based on availability of participants and to avoid any delay in treatment receipt.
  Interventions: Behavioral: Stimulus Control Instructions and Sleep Restriction Therapy
- Sleep Restriction Therapy (SRT) (Experimental): SRT aims at consolidating sleep by limiting sleep to a specified time and restricting the amount of time spent in bed. Sleep time is individualized based on the persons' sleep needs, and the sleep-wake schedule is planned to fit the persons' lifestyle. The sleep-wake schedule is changed to accommodate improvements in the persons' sleep, over time.. A trained therapist will deliver the session in which the following topics will be covered: education about sleep, factors that influence sleep, behaviors that promote or interfere with sleep, and SRT. The session will be offered in a small group (4-6) format, based on availability of participants and to avoid any delay in treatment receipt.
  Interventions: Behavioral: Stimulus Control Instructions and Sleep Restriction Therapy
- No therapy (No Intervention): No behavioral therapy for the management of insomnia is provided. However, a list of general recommendations and suggestions are provided to participants.

INTERVENTIONS:
Behavioral: Stimulus Control Instructions and Sleep Restriction Therapy — Please refer to arm/group descriptions.
  Arms: Sleep Restriction Therapy (SRT); Stimulus Control Instructions (SCI)

SUMMARY:
Research has shown that persons who have trouble sleeping and experience stress are at risk of developing heart diseases. Two treatments, called stimulus control instructions and sleep efficiency treatment, that do not involve sleeping pills, have been found effective in managing trouble sleeping. This study will be undertaken to find out if the two treatments are effective in improving sleep, and reducing stress and the risk of heart diseases. Persons with trouble sleeping may have a preference for either treatment. It is believed that if persons get the treatment they prefer, then they will be satisfied with the treatment and comply with it, and experience improvement in their sleep. This study will also examine the extent to which giving persons the treatment of their choice, as compared to giving persons treatment based on chance, will lead to higher satisfaction and compliance with treatment, and improved sleep. About 300 persons who experience trouble sleeping will be included in the study. They will be requested to complete a questionnaire and a sleep diary before and after they receive treatment, as well as 6 month and one year later.

DETAILED DESCRIPTION:
Background and Significance: Accumulating evidence indicates that sleep quantity (low number of sleep hours) and quality (subjective complaint of insomnia) are associated with an increased risk of cardiovascular diseases even after controlling for other cardiovascular risk factors. The prevalence of insomnia increases with age. Assisting middle-aged and older adults manage insomnia is essential to promote sleep, reduce anxiety and depression, and reduce the risk of cardiovascular diseases. Two behavioral treatments, stimulus control instructions (SCI) and sleep restriction therapy (SRT) are established treatments for insomnia. However, both treatments demand commitment to changing one's habits and lifestyle. Preferences for treatment have been found to influence adherence to, and outcomes of treatment. The study will provide experimental evidence of the extent to which improved sleep quantity and quality reduce the risk of cardiovascular diseases, and the SCI and SRT are effective in achieving these outcomes. The study is the first to examine satisfaction with treatment as the mechanism mediating the influence of preferences on treatment adherence and outcomes.

Objectives: The study addresses substantive and methodological areas of interest to the funding opportunity. The substantive objectives are: 1) to examine the direct effects of SCI and SRT on sleep (quantity and quality), psychological (anxiety, depression), and physical (cardiovascular symptoms and events) outcomes, and 2) to examine the indirect effects of SCI and SRT on psychological and physical outcomes, mediated through sleep quantity and quality. The methodological objectives are: 1) to compare participants randomized to treatment and participants allocated to treatment of choice on attrition, satisfaction with treatment, adherence to treatment, and sleep, psychological and physical outcomes; 2) among randomized participants, to compare those who receive and those who do not receive the preferred treatment on attrition, satisfaction with, and adherence to treatment, and sleep, psychological, and physical outcomes; and, 3) to explore the extent to which satisfaction with treatment mediates the influence of preferences on treatment adherence and outcomes.

Design: A two-stage partially randomized clinical trial will be used. Eligible participants will be randomized to the random and preference arms of the trial. In the random arm, participants will be randomly assigned to no-treatment, SCI or SRT. In the preference arm, participants will be allocated to SCI or SRT based on their preferences. Outcome data will be collected at 4 time points: pretest, posttest, and 6-month and 12-month follow-up.

Sample: Non-institutionalized, cognitively intact, adults (> 40 years) will be included if they complain of difficulty initiating and/or maintaining sleep (> 30 minutes per night, for > 3 nights per week, for > 6 weeks) that is not associated with sleep apnea. A sample of 60 participants per group, for a total of 300, is required to detect medium effects of the behavioral treatments and treatment preferences on sleep outcomes.

Measures: All outcomes will be measured with established measures. Adherence to treatment will be estimated with relevant data from the daily sleep diary. Preferences for, and satisfaction with treatment will be assessed with self-report instruments developed by the investigators and found reliable.

Analysis: In addition to descriptive statistics, hierarchical linear models and latent growth curve modeling will be used to address the objectives. The analysis will be repeated for participants who did and did not report cardiovascular diseases at baseline.

ELIGIBILITY:
Inclusion Criteria:

Persons with insomnia will be eligible for the study if they:

1. are community-dwelling, non-institutionalized middle-aged or older adults (> 40 years of age),
2. have the ability to read and write English (required for providing written consent), and
3. complain of difficulty initiating and/or maintaining sleep, manifested in sleep onset latency and/or time awake after sleep onset of 30 minutes or more per night, for a minimum of 3 nights per week, for a duration of at least 6 weeks (NIH, 2005), ascertained with relevant questions of the Insomnia Interview Schedule (Morin, 1993).

Persons with insomnia will be selected if their insomnia is primary (i.e., not related to any other condition), or comorbid associated with pre-existing cardiovascular disease, anxiety, and depression only.

Exclusion Criteria:

1. cognitive impairment as ascertained by the Mini-Mental State Exam (MMSE) score < 24 (Crum et al., 1993); cognitive impairment interferes with participants' understanding of, and ability to implement the behavioral interventions; and
2. confirmed medical diagnosis and current treatment for sleep apnea as reported by participants; SCI and SRT are not recommended for sleep apnea.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2009-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Sleep Outcome Sleep Quantity Change over time | Sleep Quantity data will be collected at 4 time points: approximately at 2 weeks (pretest), posttest (at 5 weeks), 6-month and 12-month (1 year)
  Sleep Outcomes include: sleep duration, sleep onset latency, wake after sleep onset, sleep efficiency, and daytime fatigue. The daily sleep diary (DSD) will be completed by participants to assess sleep quantity. The DSD is a self-administered log of nightly sleep behaviors. The DSD was developed by Morin (1993).
Sleep Outcome: Sleep Quality change over time | Sleep Quality data will be collected at 4 time points: at 2 weeks (pretest), posttest (at 5 weeks), 6-month and 12-month (1 year)
  Insomnia Severity Index (ISI)

SECONDARY OUTCOMES:
Psychological Outcomes: Anxiety change over time | Psychological Outcome data will be collected at 4 time points: at 2 weeks (pretest), posttest (at 5 weeks), 6-month and 12-month (1 year)
  Anxiety will be assessed with the 20-item State Trait Anxiety Inventory (STAI).
Psychological Outcomes: Depression change over time | Psychological Outcome data will be collected at 4 time points: at 2 weeks (pretest), posttest (at 5 weeks), 6-month and 12-month (1 year)
  Center for Epidemiology Studies - Depression (CESD) scale
Physical Outcomes: Cardiovascular Symptoms and Events Change over time | Physical Outcome data will be collected at 4 time points: at 2 weeks (pretest), posttest (at 5 weeks), and 6-month and 12-month follow-up (1 year).
  Physical outcomes include: cardiovascular symptoms and self-reported occurrence of cardiovascular events. The cardiovascular symptoms of chest pain, dyspnea, presyncope, and palpitation will be measured with relevant items derived from the Symptom Checklist (SCL) - 90R.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Souraya Sidani, PhD, Principal Investigator — Toronto Metropolitan University

REFERENCES:
- [Result] Ibrahim S, Sidani S. Preferences for behavioral therapies for chronic insomnia. Health 5(11): 1784-1790, 2013.
- [Derived] Sidani S, Fox M, Streiner DL, Miranda J, Fredericks S, Epstein DR. Examining the influence of treatment preferences on attrition, adherence and outcomes: a protocol for a two-stage partially randomized trial. BMC Nurs. 2015 Nov 9;14:57. doi: 10.1186/s12912-015-0108-4. eCollection 2015. PMID 26557787
- See also: Related Info — http://file.scirp.org/Html/7-8202490_39459.htm